CLINICAL TRIAL: NCT02343744
Title: A Phase 3, Multicenter, Open-Label Study Evaluating the Efficacy and Safety of CNTO1959 (Guselkumab) in the Treatment of Subjects With Generalized Pustular Psoriasis or Erythrodermic Psoriasis
Brief Title: An Efficacy and Safety Study of CNTO1959 (Guselkumab) in the Treatment of Participants With Generalized Pustular Psoriasis or Erythrodermic Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR104128; CNTO1959PSO3005 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Pustular Psoriasis
Keywords: Generalized Pustular Psoriasis; Erythrodermic Psoriasis; Guselkumab; CNTO1959
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Guselkumab (Experimental): Participants will receive 50 milligram (mg) guselkumab subcutaneously at Weeks 0, 4 and 12. At Week 16 through the study end (Week 52) participants who are defined "Very much improved" or "Much improved" in Clinical Global Impression (CGI) will continue to receive guselkumab 50 mg every 8 weeks from Week 20 to the study end (Week 52). At each visit timing from Week 20, participants who are defined "No change" or "Worsened" in CGI will receive guselkumab 100 mg and continue 100 mg every 8 weeks dosing until the study end (Week 52). Participants who are defined "Minimally improved" in CGI will also receive guselkumab 100 mg only if the investigator considers that it is necessary.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Participants will receive 50 milligram (mg) guselkumab subcutaneously at Weeks 0, 4 and 12. At Week 16 through the study end (Week 52) participants who are defined "Very much improved" or "Much improved" in Clinical Global Impression (CGI) will continue to receive guselkumab 50 mg every 8 weeks from Week 20 to the study end (Week 52). At each visit timing from Week 20, participants who are defined "No change" or "Worsened" in CGI will receive guselkumab 100 mg and continue 100 mg every 8 weeks dosing until the study end (Week 52). Participants who are defined "Minimally improved" in CGI will also receive guselkumab 100 mg only if the investigator considers that it is necessary.
  Other Names: CNTO 1959

SUMMARY:
The purpose of this study is to examine descriptively the efficacy of CNTO 1959 in participants with generalized pustular psoriasis (GPP) or erythrodermic psoriasis (EP).

DETAILED DESCRIPTION:
This is a phase 3, multicenter (when more than one hospital or medical school team work on a medical research study), open-label study evaluating the efficacy and safety of CNTO1959 (Guselkumab) in the treatment of participants with GPP or EP. Participants will receive 50 milligram (mg) guselkumab subcutaneously at Weeks 0, 4 and 12. At Week 16 up to Week 52 participants who will be defined "Very much improved" or "Much improved" in Clinical Global Impression (CGI) will continue to receive guselkumab 50 mg every 8 weeks from Week 20 to the study end (Week 52). At each visit timing from Week 20, participants who will be defined "No change" or "Worsened" will receive guselkumab 100 mg and continue 100 mg every 8 weeks dosing until Week 52. Participants who are "Minimally improved" will also receive guselkumab 100 mg only if investigator considers it necessary. Participants will primarily be assessed for the treatment success. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of generalized pustular psoriasis (GPP) or erythrodermic psoriasis (EP) at screening. A diagnosis of GPP must be classified on the basis of the criteria for diagnosis of GPP by Japanese Dermatological Association (JDA)
* Have a history of plaque-type psoriasis if subjects have a diagnosis of EP
* Have an involved body surface area (BSA) of lesion greater than or equal to (>=) 80 percent (%) at baseline if subjects have a diagnosis of EP.
* Be a candidate for phototherapy or systemic treatment for psoriasis (either naïve or history of previous treatment)
* Before the first administration of study drug, a woman must be either not of childbearing potential or of childbearing potential and practicing a highly effective methods of birth control, consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies

Exclusion Criteria:

* Has a total score of JDA severity index for GPP >=14 at baseline if subjects have a diagnosis of GPP
* Has a differential diagnosis of the erythroderma (exmaple (eg), erythroderma caused by lymphoma or drug eruption) other than EP.
* Has refused hospitalization though the investigator needed hospitalization
* Has body mass index (BMI) less than (<) 18 kilogram per square meters (kg/m^2) or meets the following modified criteria for cachexia.
* Has a BMI < 20 kg/m^2 and has lost more than 5% of their body weight in the previous months, and 4 out of the following are present: a) decreased muscle strength b) fatigue or reduced physical activity c) anorexia d) low muscle mass e) CRP greater than (>) 7 mg/L 6) hemoglobin (Hb) <12 gram per deciliters (g/dL) f) serum albumin < 3.0 g/dL
* Has Common Terminology Criteria for Adverse Events (CTCAE) Version 4 Grade 2 or higher heart failure or CTCAE v.4 Grade 3 or higher kidney failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2015-12-04 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment Success at Week16 | Week 16
  Treatment success is defined as "Very much improved", "Much improved" or "Minimally improved" in Clinical Global Impression (CGI) scale. The CGI scale is a brief clinician-rated instrument which has five categories (Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Worsened (5).

SECONDARY OUTCOMES:
Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 16 and Over Time | Baseline, Week 16, 28, 36, 48 and 52
  Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. A score less than (<) 6 indicates that psoriasis has small or no effect at all on participant's life. In addition to evaluating overall quality of life (QOL) can be used to assess 6 different aspects that may affect QOL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment.
Percentage of Participants with Treatment Success Over Time | Baseline and Every 4 weeks up to Week 52
  Treatment success is defined as "Very much improved", "Much improved" or "Minimally improved" in Clinical Global Impression (CGI) scale. The CGI scale is a brief clinician-rated instrument which has five categories (Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Worsened (5).
Percentage of Participants With Investigator's global assessment (IGA) score of 0 or 1 at Week 16 and over time | Week 16, 28, 36, 48 and 52
  Investigator's global assessment (IGA) score is Investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Percent Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 16 and over time | Week 16, 28, 36, 48 and 52
  The Psoriasis Area and Severity Index (PASI) is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a total numeric score that can range from 0 to 72.
Change From Baseline in Total and Component Japanese Dermatological Association (JDA) Severity Index for Generalized Pustular Psoriasis (GPP) Over Time | Baseline, Week 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, 48 and 52
  Japanese Dermatological Association (JDA) severity index for GPP consists of area of etythema with pustules, area of erythema (total), area of edema, fever, white blood cells (WBC), high sensitivity C-reactive protein (hsCRP) and serum albumin. The total score of JDA severity index for GPP is assigned a score of 0-17 (0=best, 17=worst).
Change From Baseline in Components of the JDA Severity Index for GPP Over Time | Baseline, Week 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, 48 and 52
  Area of erythema with pustules, area of erythema (total), area of edema are rated as 0 to 3. Fever, WBC, hsCRP and serum albumin are rated as 0 to 2.
Change From Baseline in Observed Value of Components of the JDA Severity Index for GPP Over Time | Baseline, Week 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, 48 and 52
  Area of erythema with pustules, area of erythema (total), area of edema are rated as 0 to 3. Fever, WBC, hsCRP and serum albumin are rated as 0 to 2.
Change From Baseline in Body Surface Area (BSA) of Involvement of Lesion for Erythrodermic Psoriasis (EP) Over Time | Baseline, Week 1, 2, 4, 6, 8, 16, 28, 36, 48 and 52
  Calculation of BSA involvement in dermatological lesion is used to measure disease severity and treatment responses for participants with EP.
Percentage of Participants with DLQI Score of 0 or 1 Over Time in Participants With Baseline DLQI More Than 1 | Baseline, Week 8, 16, 28, 36, 48 and 52
  Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. A score less than (<) 6 indicates that psoriasis has small or no effect at all on participant's life. In addition to evaluating overall quality of life (QOL) can be used to assess 6 different aspects that may affect QOL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment.
Percentage of Participants With a Reduction of 5 or More Points in DLQI Score Over Time | Baseline, Week 8, 16, 28, 36, 48 and 52
  Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. A score less than (<) 6 indicates that psoriasis has small or no effect at all on participant's life. In addition to evaluating overall quality of life (QOL) can be used to assess 6 different aspects that may affect QOL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment.
Change From Baseline in Physical and Mental Component Summary Scores of SF-36 Over Time | Baseline, Week 16, 28, 36 and 48
  The Short Form Health Survey (SF-36) is a generic 36-item questionnaire measuring health-related quality of life (HRQL) having 2 measures: physical component summary (PCS) and mental component summary (MCS). It consists of 8 subscales. The PCS is represented by 4 subscales: physical function, role limitations due to physical problems, pain, and general health perception. The MCS is represented by 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; zero= worst HRQL, 100=best HRQL. PCS and MCS scores are constructed as a T-score with a mean of 50 and standard deviation of 10 and no minimum or maximum score; higher scores indicate better health status.
Change From Baseline in Work Productivity and Activity Impairment (WPAI): Psoriasis (PSO) Over Time | Baseline, Week 16, 28, 36 and 48
  Work productivity was measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). The WPAI questionnaire is used to measure productivity loss associated with psoriasis during the past 7 days. It consists of six questions about absence from work because of psoriasis, hours actually worked, reduction in productivity at work attributed to psoriasis and reduction in productivity while performing daily activities. This instrument generates four scores between 0 and 100: absenteeism (work time missed), presenteeism (impairment at work / reduced productivity while working), work productivity loss (overall work impairment /absenteeism plus presenteeism) and activity impairment, which were expressed in percentage of impairment.
Observed Serum Guselkumab Concentrations | Baseline, Pre-dose on Week 4, 8, 12, 16, 20, 24, 28, 36, 44, 48 and 52
Number of Participants With Guselkumab Antibodies | Baseline, Pre-dose on Week 4, 16, 28, 48 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (20):
- Japan (20):
  - Asahikawa
  - Fukuoka
  - Gifu
  - Izumo
  - Kawasaki
  - Kita-Gun
  - Kochi
  - Kurume
  - Matsumoto
  - Miyagi
  - Morioka
  - Nagoya
  - Sapporo
  - Shimotsuke
  - Tokushima
  - Tokyo
  - Tsu
  - Tsukuba
  - Ube
  - Yokosuka